CLINICAL TRIAL: NCT02208232
Title: Observation of Rotation of the MC 6125 AS Intraocular Lens
Brief Title: Observation of Rotation of an Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Ao.Univ.-Prof. Dr.med.univ., Medical University of Vienna
Other Study IDs: EK Nr: 1267/2012
Record Dates: First submitted 2014-03-27; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Cataract
Keywords: IOL rotation
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

GROUPS / COHORTS (1):
- MC 6125 AS IOL: cataract surgery with implantation of intraocular lens MC 6125 AS in one eye
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — cataract surgery with implantation of intraocular lens

SUMMARY:
The purpose of this study is to assess the axial IOL rotation after surgery with an MC 6125 AS IOL.

At the end of surgery the orientation of the IOL is documented with a short video clip via the operating microscope unit. Follow-up examinations are performed 1 hour, 1 week and 6 months after surgery. Rotational stability of the IOL is assessed using retroillumination images with a method to avoid bias from cyclorotation or head tilt.

ELIGIBILITY:
Inclusion Criteria:

* Uni or bilateral age-related cataract necessitating phacoemulsification extraction and posterior IOL implantation

Exclusion Criteria:

* Preceding ocular surgery or trauma
* Recurrent intraocular inflammation of unknown etiology
* Uncontrolled glaucoma
* Uncontrolled systemic or ocular disease
* Blind fellow eye
* Microphthalmus
* Corneal abnormality
* History of uveitis/iritis
* Iris neovascularization
* Pseudoexfoliation
* Proliferative diabetic retinopathy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eyes of patients with uni- or bilateral cataract applying for cataract surgery at the Department of Ophthalmology, Medical University Vienna.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
IOL rotation | 6 months
  The rotation of the IOLs over the first 6 postoperative months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology and Optometry of the Medical University Vienna, Vienna, Vienna, Austria